CLINICAL TRIAL: NCT00540046
Title: Immediate vs. Delayed Post-abortal Copper T 380A IUD Insertion in Cases Over 12 Weeks of Gestation
Brief Title: Immediate vs. Delayed Insertion of Copper T 380A IUD After Termination of Pregnancy Over 12-weeks Gestation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Miriam Cremer, Clinical Assistant Professor, NYU Langone Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Post Abortion Copper T IUD
Record Dates: First submitted 2007-10-04; First posted 2007-10-05 (Estimated); Results first posted 2015-01-13 (Estimated); Last update posted 2015-02-09 (Estimated); Status verified 2015-01

CONDITIONS: Contraception Behavior
Keywords: IUD; Second trimester termination; Contraception
MeSH Terms: conditions — Contraception Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A/Immediate (Active Comparator): The patients in the immediate arm will have the Copper T 380A IUD inserted within 15 minutes after delivery of the placenta immediately following procedure
  Interventions: Device: Copper T 380A IUD
- B/Delayed (Active Comparator): The delayed group will have the Copper T 380A IUD inserted at the post-operative visit within 2-4 weeks following the procedure.
  Interventions: Device: Copper T 380A IUD

INTERVENTIONS:
Device: Copper T 380A IUD — Copper T 380A IUD will be placed at the 2-4 week post-operative visit.

SUMMARY:
The purpose of this study is to compare delayed vs. immediate insertion of the Copper T 380 IUD after termination of pregnancy after 12 weeks.

DETAILED DESCRIPTION:
Patients presenting to ParkMed Women's Clinic and the Reproductive Choice clinic at Bellevue Hospital for second trimester termination will be offered participation in this study. They will be randomized to either delayed or immediate Copper T 380A IUD insertion. The subjects will be seen at a 6 month follow-up visit and Copper T 380A IUD placement will be verified by physical exam. At this 6 month follow-up visit, subjects will fill out a satisfaction questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* women 16 years of age and older
* intrauterine pregnancy > 14 weeks gestation
* desires termination of pregnancy
* desires IUD for contraception
* ability to give informed consent
* no contraindication for D+E

Exclusion Criteria:

* unable to give informed consent
* less than 16 years of age
* congenital or acquired uterine anomaly including fibroids if they distort the uterine cavity
* acute pelvic inflammatory disease (PID)
* known or suspected uterine or cervical neoplasia or unresolved abnormal PAP smear
* untreated acute cervicitis or vaginitis, until infection treated/controlled
* confirmed Chlamydia trachomatis or Neisseria gonorrhea infection in the previous 90 days
* acute liver disease or liver tumor (benign or malignant)
* woman or partner currently with multiple sexual partners
* history of Wilson's disease
* hypersensitivity to any component of Copper T IUD

Min Age: 16 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 215 (Actual)
Dates: Start 2007-04; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Miriam L. Cremer, MD, MPH, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (2):
- United States (2):
  - Bellevue Hospital, New York, New York
  - Parkmed Women's Clinic, New York, New York

RESULTS

PARTICIPANT FLOW:
Groups:
- A/Immediate: The patients in the immediate arm will have the Copper T 380A IUD inserted within 15 minutes after delivery of the placenta immediately following procedure
  Copper T 380A IUD: Copper T 380A IUD will be placed immediately following the procedure.
Period: Overall Study
Arm/Group | A/Immediate | B/Delayed
Started | 104 | 111
Completed | 71 | 88
Not Completed | 33 | 23
Not completed — Lost to Follow-up | 33 | 23

BASELINE CHARACTERISTICS:
Population: 215 subjects were enrolled and randomized to the A/Immediate or B/Delayed group.
Groups:
- Total: Total of all reporting groups
Arm/Group | A/Immediate | B/Delayed | Total
Number analyzed (Participants) | 104 | 111 | 215
Age, Continuous [Mean (Full Range); unit: years] | 24 [16 to 41] | 23.4 [16 to 43] | 23.7 [16 to 43]
Sex/Gender, Customized [Number; unit: participants]
  Female | 104 | 111 | 215
Race/Ethnicity, Customized [Number; unit: participants]
  Black | 48 | 52 | 100
  Hispanic or Latino | 43 | 39 | 82
  White | 4 | 6 | 10
  Asian or South Asian | 1 | 4 | 5
  Mixed | 4 | 5 | 9
  Other | 2 | 3 | 5
  Missing | 2 | 2 | 4
Gestational age [Mean (Full Range); unit: weeks] | 19.2 [12 to 24] | 18.8 [12 to 24] | 19.0 [12 to 24]

OUTCOME MEASURES:

1. Primary Outcome: Use of IUD
Description: Number of participants using Copper T380A IUD 6 months after surgery
Time Frame: 6 months
Measure: Number; unit: participants
Arm/Group | A/Immediate | B/Delayed
Number analyzed (Participants) | 71 | 88
participants | 58 | 25

2. Secondary Outcome: Expulsion
Description: IUD was not removed by provider but fell out on its own.
Time Frame: 6 months
Population: The analysis here includes the 64/71 A/Immediate arm and 26/88 B/Delayed arm who received an IUD. In the A/Immediate arm, 5 women changed their mind post-randomization and in 2 cases, the provider chose not to place it. In the B/Delayed arm, reasons included not returning for follow-up visit, changing mind, and provider not wanting to place IUD.
Measure: Number; unit: percentage of expulsions
Groups:
- A/Immediate: The patients in the immediate arm had the Copper T 380A IUD inserted within 15 minutes after delivery of the placenta immediately following procedure.
  IUD status was known six months post-abortion and insertion.
- B/Delayed: The delayed group had the Copper T 380A IUD inserted at the post-operative visit within 2-4 weeks following the procedure.
  IUD status was known six months post-abortion.
Arm/Group | A/Immediate | B/Delayed
Number analyzed (Participants) | 64 | 26
percentage of expulsions | 3.1 | 0

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | A/Immediate | B/Delayed
Serious Adverse Events (participants affected / at risk) | 0/104 | 0/111
Other Adverse Events (participants affected / at risk) | 2/104 | 0/111
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | A/Immediate (N=104) | B/Delayed (N=111)
Expulsion (Reproductive system and breast disorders) | 2 (2) | 0 (0)

LIMITATIONS AND CAVEATS:
IUD presence not always confirmed by a provider at 6-month visit but self-reported.

Study not powered to detect a difference in expulsion rates due to prohibitively high sample size.

Very high-risk population.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No